CLINICAL TRIAL: NCT01856660
Title: Bitter Taste Phenotype as an Adjunct to Behavioral Weight-loss Intervention in Women
Brief Title: Bitter Taste and Weight Loss in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Beverly J Tepper, Ph.D., PhD, Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHA12060259
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss; Body Weight Change; Taste; Taste Phenotype; Lifestyle Intervention
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight Changes | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Fat Diet (Experimental): Participants are provided with a 6-month standard lifestyle intervention. They will follow an energy restricted, low-fat diet where the daily energy consumption target is 1,200- 1,500 kilocalories/d. The fat intake target is 28% or less of daily kilocalories. Gradual increase in physical activity until participants are active at least 40 min per day, 5 times/week.
  Interventions: Behavioral: Low-fat Diet
- Low-Carbohydrate Diet (Experimental): Participants are provided with a 6-month standard lifestyle intervention. They will follow a low-carbohydrate diet where the daily carbohydrate target is 50g/d. There is no energy restriction. Gradual increase in physical activity until participants are active at least 40 min per day, 5 times/week.
  Interventions: Behavioral: Low-Carbohydrate Diet

INTERVENTIONS:
Behavioral: Low-Carbohydrate Diet — Participants are provided with a 6-month standard lifestyle intervention where carbohydrate intake is limited to 50 g/day. There is no calorie restriction for participants following the Low-Carbohydrate diet. Gradual increase in physical activity across the trial to > 40 min per day, 5 times/week.
  Arms: Low-Carbohydrate Diet
Behavioral: Low-fat Diet — Participants are provided with a 6-month standard lifestyle intervention. They will follow an energy restricted, low-fat diet where the daily energy consumption target is 1,200- 1,500 kilocalories/d. The fat intake target is 28% or less of daily kilocalories. Gradual increase in physical activity until participants are active at least 40 min per day, 5 times/week.
  Arms: Low-Fat Diet

SUMMARY:
Individual food preferences are not considered in designing weight-loss therapies. This project will determine if short-term weight-loss is improved by matching participants with diets that reflect their genetically-determined food preferences.

DETAILED DESCRIPTION:
Dislike of the diet is a common complaint in weight loss therapy that contributes to poor outcomes. Ironically, individual food preferences are rarely taken into account in designing weight-loss interventions. In the proposed research, we will utilize genetically-determined differences in food preferences, indexed by PROP bitter taste phenotype to develop a novel approach to weight loss therapy. The overall goal of this project is to determine if weight loss following a 6 month intervention can be substantially improved by matching participants with diets that reflect their genetically-determined food preferences. The study is designed as a randomized clinical weight-loss intervention trial in women in which PROP non-tasters and super-tasters. will be randomized to either the low-carbohydrate or the low-fat diet condition

ELIGIBILITY:
Inclusion Criteria:

Body mass index (BMI) between 27 and 40 kg/m squared No weight loss for 3 months prior to the study Stable hypertension, dyslipemia or Type 2 diabetes - with permission from primary care provider Oral therapy to treat Type 2 diabetes - with permission from primary care provider.

Able to walk 2 block without stopping

Exclusion Criteria:

Pregnant, lactating or planning to become pregnant during the trial History of cardiovascular disease (infarct, angina, arrhythmia or stroke) Recent chemotherapy or radiation therapy Liver, renal or thyroid disease Concurrent or recent (last 6 months) participation in any other weight loss intervention Insulin injection Medications to control appetite or weight Major psychiatric illnesses

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 0, 3 months, and 6 months
  Change in weight (Kg)

SECONDARY OUTCOMES:
Diet | 0, 3 months, and 6 months
  4-day diet records will be assessed for kilocalories and macronutrients

OTHER OUTCOMES:
Physical Activity | 0, 3 months, and 6 months
  Physical activity energy expenditure will be assessed by activity monitor
Eating Attitudes | 0, 3 months, and 6 months
  Eating attitudes will be assessed with the Three-Factor Eating Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Beverly J Tepper, PhD, Principal Investigator — Rutgers University, Deptartment of Food Science
Locations (1):
- Rutgers University, Department of Food Science, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Burgess B, Raynor HA, Tepper BJ. PROP Nontaster Women Lose More Weight Following a Low-Carbohydrate Versus a Low-Fat Diet in a Randomized Controlled Trial. Obesity (Silver Spring). 2017 Oct;25(10):1682-1690. doi: 10.1002/oby.21951. Epub 2017 Aug 25. PMID 28841772
- [Derived] Burgess B, Rao SP, Tepper BJ. Changes in liking for sweet and fatty foods following weight loss in women are related to prop phenotype but not to diet. Obesity (Silver Spring). 2016 Sep;24(9):1867-73. doi: 10.1002/oby.21570. Epub 2016 Jul 19. PMID 27430708